CLINICAL TRIAL: NCT07100275
Title: The Effect of Video-Supported Online Preoperative Education on Fear, Anxiety, Sleep, and Stress in Patients Undergoing Laparoscopic Cholecystectomy: A Randomised Controlled Trial
Brief Title: The Effect of Video-Supported Online Preoperative Education on Fear, Anxiety, Sleep, and Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bingol University (Other)
Responsible Party: Principal Investigator, Izzettin Ekinci, INSTRUCTOR, Bingol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BU-SHMYO-IE-01
Record Dates: First submitted 2025-06-18; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Patient Education; Surgical Fear and Worrying; Surgical Stress Response; Medical-surgical Nursing
Keywords: Laparoscopic cholecystectomy; Preoperative education; Preoperative anxiety; Surgical fear; Sleep quality; Stress levels
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: two-group randomized controlled trial
Who Masked: Participant
Masking Description: Patients whose eligibility for the study is assessed will be stratified as male and female and then randomly assigned to two groups, the study and control groups, in a blinded manner, using the randomizer org. computer program (https://randomizer.org/).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Clinical Care (No Intervention): Control Group
- Follow-up via Mobile Health Application (Experimental): Intervention Group
  Interventions: Behavioral: Patient education; Behavioral: Follow-up via Mobile Health Application

INTERVENTIONS:
Behavioral: Patient education — In addition to the procedures in the control group, the patient will be informed about the surgery while he/she is at home the day before the surgery. Information will be provided about the hospital and surgical process. If there are any questions, the patient will be asked and their concerns will be resolved. T0-T1-T2 procedures will be performed on patients in the intervention group, respectively.
  Other Names: Online video-assisted patient education; Surgical fear and anxiety
  Arms: Follow-up via Mobile Health Application
Behavioral: Follow-up via Mobile Health Application — The researcher will create a video depicting the process of transferring patients from the ward to surgery. The video will be created with a volunteer mannequin. It will not be created with a real patient. This video will be recorded during a non-busy Sunday at the hospital. This video will be shown to patients the evening before surgery, following online education, and their questions will be answered.
  Arms: Follow-up via Mobile Health Application

SUMMARY:
Gallbladder stone disease is among the most common digestive system problems worldwide. The global incidence of gallstones is estimated to be 10-20%. In Europe, this rate is approximately 20%. In Turkey, the incidence of gallstones is accepted as 6% and it is estimated that an average of 4 million people have gallstones. ). Laparoscopic cholecystectomy is the most commonly used minimally invasive technique in the surgical treatment of gallbladder diseases. Although this is a technique, it also has many complications. Although drains placed after surgery are protective and therapeutic, they may cause some complications. Due to all these reasons, there are disadvantages such as lack of training and incomplete information given to the patient before surgery, and the patient not knowing what to do in physiological and psychological preparation before surgery. This training and information seems to be important in post-operative recovery and shortening the hospital period. Pre-surgical virtual training enables early detection of changes in the patient's vital signs, early intervention, and reduction of the number of home visits.

DETAILED DESCRIPTION:
This study aims to examine the effect of online education given preoperatively to patients undergoing laparoscopic cholecystectomy surgery on fear, anxiety, sleep and stress.

This randomized controlled trial will be carried out in Bingöl State Hospital Surgical Service between 2024-2025. The research population consists of patients who underwent Laparoscopic Cholecystectomy surgery in this hospital between the specified dates.

will create. The research sample will consist of 128 patients who voluntarily participate in the research.

The data to be used in the research consists of the patients' introductory information form, clinical information and survey results, and a number of tests to be measured by taking blood. While demographic information includes basic information such as age, gender, marital status and educational status, clinical information includes details about the patient's preoperative process. Survey data includes evaluations of fear, anxiety and sleep, and blood tests include serum cortisol level and serum glucose level.

The collected data will be analyzed in the SPSS statistical analysis program. In statistical analyses, methods such as descriptive statistics, t-test, ANOV will be used and relationship-seeking analyzes will be conducted on the factors affecting stress formation.

This research aims to determine the effect of online education applied to prevent fear, anxiety and stress before laparoscopic cholecystectomy surgery. The positive effects of preoperative online education on patients, whether it reduces fear, anxiety and stress, and its effects on the patient's general well-being will be evaluated.

This study, which investigates the effect of online education applied to prevent fear, anxiety and stress before laparoscopic cholecystectomy surgery, aims to make a significant contribution to the literature in this field. The findings may contribute to more effective and holistic online patient education before laparoscopic cholecystectomy surgery.

In this project, a multidisciplinary approach has been adopted and members of the team from different areas of expertise will contribute according to their areas of expertise at different stages of the project. This is critical to the successful completion of the project.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18,
* Those who can speak and write Turkish (education level primary school and above),
* Those who have undergone laparoscopic cholecystectomy surgery for the first time,
* Those who are not receiving psychiatric treatment or taking medication,
* Those who do not have a chronic disease,
* Those who are not taking cortisone-type medication,
* Those who have a smartphone and know how to use it,
* Patients whose anesthesia evaluation was performed 1-3 days before the surgery,
* Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Those whose surgery is canceled for any reason.
* Those who want to leave the study at any stage after volunteering to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Comparison Scale (VCS)-Anxiety | 1-2 Month
  It consists of a 10-cm-long horizontal line. The left side contains the labels "I don't have anxiety" and the right side "I feel a lot of anxiety." The VAS value is determined by measuring the distance between the leftmost end of the scale and the marked point. Values range from 0 to 10, with higher values indicating increased anxiety (Cline et al., 1992).

SECONDARY OUTCOMES:
Richard-Campbell Sleep Scale (RCS): | 1-2 Months
  Richard-Campbell Sleep Scale (RCS):
  Developed by Richard Campbell in 1987, this scale consists of six items that measure the quality and depth of sleep, duration of sleep, and the noise level in the sleep environment. As the scale score increases, so does sleep quality. The Cronbach's alpha for the scale was found to be 0.82.
Surgical Fear Scale | 1-2 Months
  This scale was developed by Theunissen and colleagues in 2014 to determine the fear level of patients undergoing elective surgery. The scale consists of eight items and is scored from 0 to 10. The total score is 0, with a minimum score of 80 and a maximum score of 80. Higher scores indicate higher levels of surgical fear. The Cronbach's alpha reliability coefficient for the scale was calculated as 0.89.

CONTACTS AND LOCATIONS:
Overall Officials: izzettin e researcher, Study Director; aynur koyuncu, Assistant Professor, Study Director — Hasan Kalyoncu University
Locations (1):
- Bingol Universty, Bingöl, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to ethical restrictions and data protection policies.

REFERENCES:
- [Result] Flores A, Hoffman HG, Navarro-Haro MV, Garcia-Palacios A, Atzori B, Le May S, Alhalabi W, Sampaio M, Fontenot MR, Mason KP. Using Immersive Virtual Reality Distraction to Reduce Fear and Anxiety before Surgery. Healthcare (Basel). 2023 Oct 9;11(19):2697. doi: 10.3390/healthcare11192697. PMID 37830734
- [Result] Maheta B, Shehabat M, Khalil R, Wen J, Karabala M, Manhas P, Niu A, Goswami C, Frezza E. The Effectiveness of Patient Education on Laparoscopic Surgery Postoperative Outcomes to Determine Whether Direct Coaching Is the Best Approach: Systematic Review of Randomized Controlled Trials. JMIR Perioper Med. 2024 Jun 27;7:e51573. doi: 10.2196/51573. PMID 38935953
- [Result] Richey AE, Hastings KG, Karius A, Segovia NA, Caruso TJ, Frick S, Rodriguez S. Virtual Reality Reduces Fear and Anxiety During Pediatric Orthopaedic Cast Room Procedures: A Randomized Controlled Trial. J Pediatr Orthop. 2022 Nov-Dec 01;42(10):600-607. doi: 10.1097/BPO.0000000000002250. Epub 2022 Aug 30. PMID 36040069
- [Result] Abbasnia F, Aghebati N, Miri HH, Etezadpour M. Effects of Patient Education and Distraction Approaches Using Virtual Reality on Pre-operative Anxiety and Post-operative Pain in Patients Undergoing Laparoscopic Cholecystectomy. Pain Manag Nurs. 2023 Jun;24(3):280-288. doi: 10.1016/j.pmn.2022.12.006. Epub 2023 Jan 17. PMID 36658058
- See also: Bingöl State Hospital — https://bingoldh.saglik.gov.tr/
- Available data/document: Study Protocol: Supervisory authority — https://bingolism.saglik.gov.tr/ — The management that gives the necessary permission in the hospital where the study will be conducted

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT07100275/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT07100275/ICF_001.pdf